CLINICAL TRIAL: NCT05518643
Title: Enhanced Recovery Program, Patient Reported Outcomes, Surgery-specific Outcomes and Stress Response After Pancreatic Surgery: A Prospective Observational Cohort Study by the Thessalic Pancreas Study Group (ThePANas).
Brief Title: Compliance With ERAS Protocol in Pancreatic Surgery, Stress Response and Outcomes
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Collaborators: IASO Thessalias (Other); Larissa University Hospital (Other)
Responsible Party: Principal Investigator, DESPOINA LIOTIRI, MD, DESAIC, PgCert HBE(UK), EDRA, MSc, PhD(c), Consultant Anaesthesiologist, University of Thessaly
Other Study IDs: 270; 31 (Other: IASO Thessalias); 47 (Other: IASO Thessalias)
Record Dates: First submitted 2022-08-21; First posted 2022-08-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: ERAS; Pancreas Cancer; Pancreas; Fistula; Delayed Gastric Emptying; Surgery-Complications; Pancreatic Hemorrhage; PROMs
Keywords: ERAS; Pancreas Cancer; PROMs; Stress response to surgery; Surgery-Complications; PLR; NLR; Quality of Life
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: ERAS protocol — ERAS protocol as described above

SUMMARY:
The purpose of this study is to evaluate the impact of compliance with enhanced recovery after surgery (ERAS) program on patient reported outcomes (PROs), surgery-specific outcomes and stress response after pancreatic surgery.

This prospective observational study will include all consecutive patients undergoing pancreatic surgery over a period of three years (2022 - 2025) at two sites, namely University General Hospital of Larissa and IASO Thessalias, in Greece. Patients will be prospectively enrolled after written informed consent. Data will be collected on patient characteristics, surgical and anaesthetic techniques, complications, and length of stay. Quality of life questionnaires will be administered to patients preoperatively, on the fith postoperative day, first follow-up after discharge, one month and six months after the operation. The stress response will be assessed by measuring the Neutrophil-Lymphocyte Ratio and Platelet-Lymphocyte Ratio (NLR and PLR) preoperatively, and on the first five postoperative days. Data will be collected on pancreatic surgery-specific complications such as delayed gastric emptying (DGE), post-pancreatectomy haemorrhage (PPH) and postoperative pancreatic fistula (POPF) formation. Anonymised data will be uploaded by the principal investigator on a protected excel spreadsheet for analysis.

DETAILED DESCRIPTION:
In this study the ERAS program is applied to patients undergoing pancreatic surgery.This is a prospective observational cohort study.The study will take place in two hospitals, the University General Hospital of Larissa (academic center), and IASO Thessalias (largest private general hospital in Thessaly). The study period is three years between May 2022 and April 2025. All patients undergoing pancreatic surgery during this period will be invited to participate in the study. Recruitment will take place at the first appointment with the surgeon when the patient is listed for surgery. The patient will be provided with detailed information about the program which also includes an information leaflet. A written consent form will be signed by patients willing to participate in the study.

Enrolled patients will follow the ERAS pathway for pancreatic surgery during the preoperative, intraoperative, and postoperative period. The ERAS protocol is based on ERAS society recommendations for enhanced recovery after pancreatoduodenectomy.

The ERAS protocol consists of the following items:

First appointment preoperative:

* Patient education about the program
* Prehabilitation with advice on physical exercise and nutritional support
* Advice to stop smoking and alcohol consumption
* Plan for optimisation of comorbidities
* Completion of quality of life questionnaire

Day before surgery:

* Discussion about the program to address any patient concerns and anxieties
* Light meal and carbohydrate drink before bedtime
* Anti-clotting injection 12 hours before surgery

Day of surgery:

* Carbohydrate drink and painkillers 3 hours before surgery
* Clear fluids allowed up to 3 hours before surgery
* Antibiotics within 1 hour before surgical incision

Intraoperative

* Epidural catheter is sited before general anaesthesia
* Multimodal and opioid-sparing analgesia
* Nausea and vomiting prophylaxis
* Goal directed fluid therapy
* Active warming to avoid hypothermia
* Monitoring of blood glucose to maintain normoglycaemia
* Bile culture
* Repeat antibiotics if surgery lasts more than 4 hours

Postoperative:

* Removal of nasogastric tube by postoperative day 1
* Removal of drains by postoperative day 3
* Multimodal analgesia, epidural catheter for 3 days, minimisation of opioids
* Early and scheduled mobilisation and respiratory physiotherapy protocol
* Diet protocol with nutritional drinks and gradual progression from light to solid diet by postoperative day 5
* Removal of urinary catheter when patients able to mobilise on their own, by postoperative day 5
* Cessation of intravenous fluids when patients able to drink 1.5 liters of water, by postoperative day 5
* Regular gastrokinetic medication and gum chewing
* Glycaemic control protocol
* Cessation of antibiotics if bile culture negative and no other indication to continue

The study group will use a checklist with ERAS criteria to follow for each patient and data will be collected on adherence rates to these criteria.

Data will be collected on patient demographics such as sex, age, Body Mass Index (BMI), American Society of Anaesthesiologists (ASA) physical status, and co-morbidities. Data will also be collected on surgical approach and technique, and tumour stage (pTNM). Data will be collected on complications including cardiovascular and respiratory complications, infectious complications (surgical site infection, chest infection, urinary tract infection, intra-abdominal abscess, sepsis), anaesthetic complications (severe pain, delirium, cognitive decline), functional complications (functional decline, new mobility aid use, pressure ulcer, discharge to nursing or rehabilitation facility), renal failure, ileus, return to theatre, readmission, and death. Data will be collected on length of stay and pancreatic surgery-specific complications such as DGE, PPH and POPF formation. International consensus guidelines will be used for definition and grading of these complications.

Quality of life will be assessed by Patient Reported Outcome Measures (PROMS). The stress response will be assessed by measuring NLR and PLR. After anonymization, all data will be prospectively uploaded by local investigators on a protected database and incorporated into a spreadsheet for data analysis.

The data will be analyzed using PROMs, NLR and PLR ratios, postoperative complications, length of hospital stay and cancer recurrence rates as the main outcome variables.The influence of the following factors will be assessed: age, BMI, sex, surgical technique, pTNM stage, preoperative comorbidity, ASA classification, previous SARS-CoV-2 infection, and compliance to the ERAS protocol (<50%, 50-70%, 70-90%, >90%). Adherence will be calculated as the number of interventions fulfilled/20 (total number of preoperative and perioperative interventions).

The statistical model will be multivariate regression analysis. Sample size guidelines for observational studies with regression analysis are based on simulation studies and suggest that the minimum number of events per variable (EPV) should be 10. According to these guidelines the minimum sample size is calculated at 90. To account for 25% loss to follow-up the investigators aim for a total enrollment goal of 120 participants. IBM® SPSS 26 software will be used for statistical analysis. Continuous variables will be compared with One-Way ANOVA or Student's t test for parametric data and with a non-parametric test (Mann-Whitney U test or Kruskal-Wallis test), as indicated. Categorical data will be analysed by using the chi squared or Fisher's exact test where indicated. Quantitative values will be expressed as mean ± standard deviation (SD), median and range, categorical data with percentage frequencies. The odds ratio (OR) will be presented followed by 95% confidence interval (95% CI). Differences in survival and complications between different degrees of compliance will be assessed by the application of log rank test. P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* all pancreatic surgery patients
* above the age of 18
* fluent greek speakers
* without communication barriers

Exclusion Criteria:

* younger than 18 years-old
* unable or unwilling to participate
* other surgical procedures
* communication barriers
* lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive community patients presented for pancreatic surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported outcomes as measured by the Health Questionnaire EORTC QLQ-C30 | 1 week to 1 day before the operation, postoperative day 5, first follow-up 1 week post discharge, 1 month, and 6 months after the operation
  This questionnaire assesses health related quality of life (HRQoL) for cancer patients and includes 30 questions. The QLQ-C30 includes five functional scales (physical, role, emotional, cognitive, and social functioning); eight symptom scales or single items (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, and diarrhea); an item to assess financial difficulties; 1 global health status scale; and 1 global quality of life scale. Each one of the first 28 items has 4 levels: 1 = not at all, 2 = a little, 3 = quite a bit, 4 = very much. The last 2 questions ask the patient to rate their own health and quality of life on a scale from 1 (very poor) to 7 (excellent). PROMs questionnaires will be distributed in paper format and filled out by pen.
Change on the stress response to surgery measured by the Neutrophil-Lymphocyte and Platelet-Lymphocyte Ratio (NLR and PLR). | 1 week to 1 day before the operation, and postoperative days 1-5
  NLR and PLR will be calculated by blood tests
Rate of Delayed Gastric Emptying (DGE) | within 6 weeks from operation
  Number of DGE defined and graded according to the International Study Group of Pancreatic Surgery (ISGPS).
Rate of Post Pancreatic Fistula (POPF) formation | within 6 weeks from operation
  Number of POPF defined and graded according to the International Study Group of Pancreatic Fistula (ISGPF).
Rate of Postoperative Pancreatic Haemorrhage (PPH) | within 6 weeks from operation
  Number of PPH defined and graded according to the International Study Group of Pancreatic Surgery (ISGPS).

SECONDARY OUTCOMES:
Length of hospital stay (LOS) | within 6 weeks from operation
  Total number of days spent in the hospital (including any readmission)
Overall morbidity rate | Within 3 months from operation
  Number of any perioperative adverse events graded according to Clavien-Dindo
Cancer recurrence rate | within 1 year from operation
  Number of patients with cancer recurrence with metastases

CONTACTS AND LOCATIONS:
Overall Officials: Despoina Liotiri, Consultant, Principal Investigator — University of Thessaly, IASO Thessalias; Dimitrios Zacharoulis, Professor, Study Chair — University of Thessaly; Eleni Arnaoutoglou, Professor, Study Director — University of Thessaly
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided
6 months after the end of the study

REFERENCES:
- [Background] Melloul E, Lassen K, Roulin D, Grass F, Perinel J, Adham M, Wellge EB, Kunzler F, Besselink MG, Asbun H, Scott MJ, Dejong CHC, Vrochides D, Aloia T, Izbicki JR, Demartines N. Guidelines for Perioperative Care for Pancreatoduodenectomy: Enhanced Recovery After Surgery (ERAS) Recommendations 2019. World J Surg. 2020 Jul;44(7):2056-2084. doi: 10.1007/s00268-020-05462-w. PMID 32161987
- [Background] Spolverato G, Maqsood H, Kim Y, Margonis G, Luo T, Ejaz A, Pawlik TM. Neutrophil-lymphocyte and platelet-lymphocyte ratio in patients after resection for hepato-pancreatico-biliary malignancies. J Surg Oncol. 2015 Jun;111(7):868-74. doi: 10.1002/jso.23900. Epub 2015 Apr 10. PMID 25865111
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Bujang MA, Sa'at N, Sidik TMITAB, Joo LC. Sample Size Guidelines for Logistic Regression from Observational Studies with Large Population: Emphasis on the Accuracy Between Statistics and Parameters Based on Real Life Clinical Data. Malays J Med Sci. 2018 Jul;25(4):122-130. doi: 10.21315/mjms2018.25.4.12. Epub 2018 Aug 30. PMID 30914854
- [Background] Austin PC, Steyerberg EW. Events per variable (EPV) and the relative performance of different strategies for estimating the out-of-sample validity of logistic regression models. Stat Methods Med Res. 2017 Apr;26(2):796-808. doi: 10.1177/0962280214558972. Epub 2014 Nov 19. PMID 25411322